CLINICAL TRIAL: NCT06842914
Title: Postural Training for Standing and Sitting in Men Suffering From Post-prostatectomy Urinary Incontinence
Acronym: EDULAPRO
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/0203/OB
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Men Who Have Undergone Prostatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: postural training — postural training

SUMMARY:
Existing research highlights the difficulty of identifying an optimal rehabilitation technique for improving male urinary continence. However, several authors have demonstrated the benefits of treatment based on improving movement control, often referred to as postural motor contro. The main principles are: respect for the neutral lumbopelvic position, reduction of intra-abdominal constraints and ecology of movement. With the aim of encouraging patient-centred clinical practice, patients are asked to fill in an assessment form on which they note the most disabling gestures with regard to their UI during the initial assessment. In our experience, 'sitting down or getting up from a chair' is the item most frequently and most severely reported. In practical terms, posture and body movements play a vital role in the management of pelvic strain. For example, excessive pressure on the bladder due to poor postural control would increase stress on the bladder. Optimal postural control would have the advantage of reducing and promoting continence mechanisms. If we take the example of the transition from sitting to standing, postural control aims to improve neuromuscular coordination and promote continence.

In the context of health education during the first session, it might be interesting to study the impact of modifying postural control when standing/sitting on urinary incontinence and how patients feel about it.

ELIGIBILITY:
Inclusion Criteria:

* Men over the age of majority.
* Men who had had a prostatectomy within one year of inclusion.
* Positive response to the question 'Do you leak urine when you stand or sit up?
* Patients with a medical prescription for post-prostatectomy urinary incontinence rehabilitation.
* Patients who are able to understand and follow the instructions relating to postural education when standing up or sitting down.
* Patients who have read and understood the information note and who have not objected to participating in the research.
* Patients affiliated to a social security scheme.

Exclusion Criteria:

* Urinary leakage before prostatectomy (diagnosed by a doctor)
* Pad test ≤ 0 grams at the inclusion visit, before showing the postural control technique.
* On anticholinergic treatment initiated less than 3 months ago.
* Impossible to carry out postural control education (spinal surgery, serious neurological or orthopaedic pathology).
* Patients deprived of their liberty by an administrative or judicial decision or protected adults (under guardianship or trusteeship).
* Participation in other interventions: Individuals participating at the same time in other post-prostatectomy rehabilitation programmes or similar clinical studies.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men who have undergone prostatectomy
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
the sign of the difference between the results of the two pad tests of 3 times 24 hours. | 15 days

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Chu Rouen, Rouen
  - Ch bretagne atlantique, Vannes

IPD SHARING:
Plan to Share IPD: No